CLINICAL TRIAL: NCT02682992
Title: A Phase II Prospective Trial of Low-Level Laser Therapy for Prevention of Oral Mucositis in Patients Receiving Chemotherapy and Radiation for Head and Neck Cancer
Brief Title: Low-Level Laser Therapy for Prevention of Oral Mucositis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: David A. Clump, MD, PhD (Other)
Responsible Party: Sponsor-Investigator, David A. Clump, MD, PhD, Assistant Professor, University of Pittsburgh
Organization: University of Pittsburgh (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 18-127
Record Dates: First submitted 2016-02-10; First posted 2016-02-17 (Estimated); Results first posted 2022-04-13 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2022-04

CONDITIONS: Mucositis
MeSH Terms: conditions — Mucositis | interventions — Low-Level Light Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Low Level Laser Therapy (Experimental): Patients meeting the eligibility criteria will be enrolled to receive prophylactic LLLT in addition to standard of care measures for oral mucositis or other toxicity of therapy. The radiation and chemotherapy dose, schedule, modality, technique, and any required adjustments will not be influenced by this protocol and will follow standard existing institutional practices.
  Interventions: Device: Low Level Laser Therapy

INTERVENTIONS:
Device: Low Level Laser Therapy — Patients will receive LLLT three times per week concurrently with chemoradiotherapy. LLLT may be delivered either immediately prior to or after the patient's daily fraction of radiotherapy. Patients will be treated extra-orally with a THOR® LED cluster for one minute along the buccal mucosa on each side and intraorally for one minute to the tongue and soft palate. During each LLLT treatment session a thorough oral exam will be performed to identify any areas of mucositis. If the patient should develop intraoral lesions they will be targeted directly with the intraoral probe for one minute to each site of mucositis. The laser settings to be used are as follows: frequency 2.5 Hz; wavelength 660 nm; and power 75 mW, for an energy of 4.5 J.

SUMMARY:
The overall purpose of this study is to examine the efficacy of prophylactic low-level laser therapy (LLLT) to reduce the incidence of oral mucositis and adverse events in patients receiving combined modality therapy consisting of chemotherapy and radiation therapy for head and neck cancer.

DETAILED DESCRIPTION:
A phase II, single-arm trial to examine the efficacy of prophylactic low-level laser therapy (LLLT) to reduce the incidence of oral mucositis and adverse events in patients receiving combined modality therapy consisting of chemotherapy and radiation therapy for head and neck cancer.

Patients meeting the eligibility criteria will be enrolled to receive prophylactic LLLT in addition to standard of care measures for oral mucositis or other toxicity of therapy. The radiation and chemotherapy dose, schedule, modality, technique, and any required adjustments will not be influenced by this protocol and will follow standard existing institutional practices.

Patients will receive LLLT three times per week concurrently with chemoradiotherapy. LLLT may be delivered either immediately prior to or after the patient's daily fraction of radiotherapy. Patients will be treated extra-orally with a THOR® LED cluster for one minute along the buccal mucosa on each side and intraorally for one minute to the tongue and soft palate. During each LLLT treatment session a thorough oral exam will be performed to identify any areas of mucositis. If the patient should develop intraoral lesions they will be targeted directly with the intraoral probe for one minute to each site of mucositis. The laser settings to be used are as follows: frequency 2.5 Hz; wavelength 660 nm; and power 75 mW, for an energy of 4.5 J.

Patients will be evaluated prior to therapy, weekly during therapy, two weeks after the completion of therapy, and three months after the completion of therapy. During each assessment, the following toxicities will be assessed: pain, mucositis, dysphagia, xerostomia, dysgeusia, dermatitis, trismus, and quality of life.

Previous studies indicate that approximately 40% of patients will experience severe mucositis with radiation and concurrent chemotherapy. The hypothesis in this trial is that the addition of LLLT to this treatment regimen will decrease the rate of severe acute OM to 20%. We plan to enroll 50 patients at our institution.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to understand and sign informed consent form approved by the HRPO.
* Males or females greater than or equal to 18 years old.
* Biopsy-proven HNC including cancers of the nasopharynx, oropharynx, larynx, hypopharynx, or HNC of unknown primary origin amenable to therapy with radiation and concurrent chemotherapy.
* Patients who are planned to receive definitive or adjuvant radiotherapy with concurrent platinum-based chemotherapy.
* Patients whose clinical treatment plans include a continuous course of external beam radiotherapy by intensity-modulated radiation therapy (IMRT) and/or image-guided radiation therapy (IGRT), given as a cumulative dose of 5000 - 7000 cGy in single daily fractions of 180 - 200 cGy, combined with a concurrent course of weekly or tri-weekly cisplatin or carboplatin chemotherapy.
* Karnofsky performance status score >60.
* Female subjects of child-bearing potential must have a negative pregnancy test prior to enrollment.

Exclusion Criteria:

* Subject has evidence of current mucositis, mucosal ulceration, or unhealed surgical wounds from surgical resection or biopsy.
* Prior radiation to the head and neck.
* Patients with gross tumor involvement of the oral cavity or oral mucosa.
* Subjects planned to receive altered fractionation radiotherapy or multiple fractions per day
* Subject is using a pre-existing feeding tube for nutritional support at the time of study entry.
* Women who are pregnant or breast-feeding.
* Subject plans to receive concurrent chemotherapy, other than the regimens specified in the inclusion criteria.
* Patients who have chronic immunosuppression or are on current immunosuppressive therapies.
* Patients who have a contraindication to radiation therapy.
* Patients enrolled on another investigational trial for oral mucositis prevention.
* Life expectancy of less than 3 months.
* Unable or unwilling to adhere to study-specified procedures

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Actual)
Dates: Start 2016-06; Primary Completion 2020-11 (Actual); Study Completion 2020-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David A Clump, MD, PhD, Principal Investigator — UPMC Department of Radiation Oncology
Locations (1):
- UPMC Shadyside Department of Radiation Oncology, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Low Level Laser Therapy: Patients that received prophylactic LLLT in addition to standard of care measures for oral mucositis or other toxicity of therapy. The radiation and chemotherapy dose, schedule, modality, technique, and any required adjustments will not be influenced by this protocol and will follow standard existing institutional practices.
  Low Level Laser Therapy: LLLT three times per week concurrently with chemoradiotherapy. LLLT may be delivered either immediately prior to or after the patient's daily fraction of radiotherapy. Patients will be treated extra-orally with a THOR® LED cluster for one minute along the buccal mucosa on each side and intraorally for one minute to the tongue and soft palate. During each LLLT treatment session a thorough oral exam performed to identify any areas of mucositis. Patients that develop intraoral lesions are targeted directly with the intraoral probe for one minute to each site of mucositis. The laser settings used are as follows: frequency 2.5 Hz; wavelength 660 nm; and power 75 mW, for an energy of 4.5 J.
Period: Overall Study
Arm/Group | Low Level Laser Therapy
Started | 47
Completed | 47
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 60.5 [54 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 41
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 40
  More than one race | 0
  Unknown or Not Reported | 2
Head Neck Origin [Count of Participants; unit: Participants]
  Hypopharynx | 1
  Larynx | 8
  Nasopharynx | 3
  Oropharynx | 33
  Unknown | 2
Tobacco History [Count of Participants; unit: Participants]
  Tobacco use - No | 25
  Tobacco use - Yes | 22
Alcohol History [Count of Participants; unit: Participants]
  Alcohol use - No | 18
  Alcohol use - Yes | 29
Positive Karnofsky Performance Status [Number; unit: participants] — Patients with a performance status score >60. The Karnofsky Performance Scale is an assessment tool of functional impairment to assess the prognosis in individual patients. The score is from 0-100%, with lower Karnofsky scores indicating the lower likelihood of survival.
  participants | 47

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Severe (WHO Grade 3-4) Oral Mucositis
Description: Percentage of participants with severe oral mucositis per the World Health Organization (WHO grade 3-4) (ulcerative lesions of the oral mucosa) in patients treated to a cumulative radiation dose of at least 5000 cGy.
Time Frame: Up to 1 year
Population: Treated patients experiencing severe oral mucositis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 23 [14.9 to 34.8]

2. Primary Outcome: Percentage of Participants With Severe (CTCAE v. 4.0 Grade 3-5) Oral Mucositis
Description: The Percentage of participants with severe Common Terminology Criteria for Adverse Events (CTCAE, v. 4.0 grade 3-5) oral mucositis in patients treated to a cumulative radiation dose of at least 5000 cGy.
Time Frame: Up to 1 year
Population: Treated patients experiencing severe oral mucositis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 23 [14.9 to 34.8]

3. Secondary Outcome: Time to Onset of Oral Mucositis
Description: Time to onset of severe oral mucositis following the initiation of radiotherapy. per Common Terminology Criteria for Adverse Events (CTCAE v. 4.0 grade 3-4) oral mucositis following the initiation of radiotherapy.
Time Frame: Up to 1 year
Population: Includes only treated patients experiencing severe oral mucositis
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 11
days | NA [NA to NA] — Median number of days and 95% Confidence Interval were not reached due to insufficient number of participants with events.

4. Secondary Outcome: Mean Cumulative Radiation Dose
Description: Mean cumulative radiation dose at time of onset of severe oral mucositis per Common Terminology Criteria for Adverse Events (CTCAE v. 4.0 grade 3-4)
Time Frame: Up to 1 year
Population: Includes only treated patients experiencing severe oral mucositis.
Measure: Mean (Standard Deviation); unit: Gy
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 11
Gy | 56 (12.8624)

5. Secondary Outcome: Duration of Oral Mucositis
Description: Time from onset of severe oral mucositis per Common Terminology Criteria for Adverse Events (CTCAE v. 4.0 grade 3-4). The duration of SOM is calculated as the time in days between the onset of SOM to the time when the patient is first found to recover from SOM. If the patient do not recover from SOM, the duration is censored at the last observation time.
Time Frame: Up to 1 year
Population: Includes only treated patients experiencing severe oral mucositis.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 11
days | 24 [14 to 89]

6. Secondary Outcome: Percentage of Participants With Feeding Tube Replacement
Description: Percentage of participants who require feeding tube placement during treatment.
Time Frame: Up to 1 year
Population: Treated patients who required feeding tube placement.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 36 [25.7 to 48.2]

7. Secondary Outcome: Percentage of Participants With Trismus
Description: Percentage of Participants with trismus (reduced opening of the jaws determined via measurement of interincisal distance). The interincisal distance will be measured in millimeters at the patient's maximum comfortable extent of mouth opening.
Time Frame: Up to 1 year
Population: Treated patients experiencing trismus.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 26 [15.3 to 39.5]

8. Secondary Outcome: Quality of Life Via Functional Assessment of Cancer Therapy Head & Neck Cancer (FACT-HN) Questionnaire
Description: This measure is based on a self-administered questionnaire. Responses to each item were on a Likert scale score ranging from 0 to 4. The individual responses were summed to compute subscale scores, and the subscales to compute overall total scores, with higher scores indicating better Quality of Life. FACT-HN includes 2 parts - FACT-G and FACT-HN. The basic FACT-G (general) is comprised of 27 items (0-108). Subscales include Physical Well-Being (0-28), Social/Family Well-Being (0-28), Emotional Well-Being (0-24), and Functional Well-Being, (0-28). Two "Relationship with physician" items (subscale score min/max = 0-8) were added to the FACT-G in this trial, for a total of 29 FACT-G items (total min/max = 0-116). The FACT-HN is comprised of 12 head and neck specific items (0-48). Thus, the overall total possible score range was 0-164. The FACT Head & Neck Trial Outcome Index is a composite score which includes only physical, functional, and FACT-HN, thus a score range from 0-104.
Time Frame: Up to 1 year
Population: Treated patients that completed Fact QoL assessments.
Measure: Median (Inter-Quartile Range); unit: score on a scale
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 36
score on a scale
  PHYSICAL WELL BEING (PWB) | 21.5417 [17.8690 to 23.875]
  SOCIAL/FAMILY WELL BEING (SWB) | 24.3654 [22.0833 to 26.7424]
  EMOTIONAL WELL BEING (EWB) | 20.9167 [18.2738 to 22.0909]
  FUNCTIONAL WELL BEING (FWB) | 18.7708 [11.6845 to 21.6307]
  FACT-G total score (FACTG) | 84.9028 [73.9515 to 92.0182]
  FACT HN | 21.7035 [18.75 to 25.6083]
  FACT-G with FACT HN total score | 107.403 [89.0835 to 117.246]
  FACT Head & Neck Trial Outcome Index | 62.4470 [46.4815 to 69.5091]

9. Secondary Outcome: Percentage of Participants With Oral Mucositis
Description: The percentage of participants with oral mucositis Common Terminology Criteria for Adverse Events (CTCAE v. 4.0 - all grades) in patients treated to a cumulative radiation dose of at least 5000 cGy.
Time Frame: Up to 1 year
Population: Treated patients experiencing oral mucositis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 96 [87.9 to 98.6]

10. Secondary Outcome: Percentage of Participants With Dysphagia
Description: Percentage of participants with dysphagia per Common Terminology Criteria for Adverse Events (CTCAE, v. 4.0) and via diet assessment.
Time Frame: Up to 1 year
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 100 [94.6 to 100]

11. Secondary Outcome: Percentage of Participants With Xerostomia
Description: Percentage of participants with xerostomia (oral dryness) per Common Terminology Criteria for Adverse Events (CTCAE) CTCAE v. 4.0.
Time Frame: Up to 1 year
Population: Treated patients experiencing xerostomia.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 100 [94.6 to 100]

12. Secondary Outcome: Percentage of Participants With Dysgeusia
Description: Percentage of participants with dysgeusia (altered taste with/without change in diet (e.g., oral supplements); noxious or unpleasant taste; loss of taste) per Common Terminology Criteria for Adverse Events (CTCAE, v. 4.0).
Time Frame: Up to 1 year
Population: Treated patients experiencing dysgeusia.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 100 [94.6 to 100]

13. Secondary Outcome: Percentage of Participants With Radiodermatitis
Description: Percentage of participants with radiodermatitis (skin response to ionizing radiation exposure/therapy ranging from erythematous rash to desquamation and necrosis) per Common Terminology Criteria for Adverse Events (CTCAE, v. 4.0).
Time Frame: Up to 1 year
Population: Treated patients experiencing radiodermatitis.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 100 [94.6 to 100]

14. Secondary Outcome: Percentage of Participants With Mouth Pain
Description: Percentage of participants with mouth pain. Mouth pain severity will be assessed using a standard 0-10 scale, with higher scores indicating greater pain.
Time Frame: Up to 1 year
Population: Treated patients experiencing mouth pain.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 94 [85.1 to 97.4]

15. Secondary Outcome: Percentage of Participants With Throat Pain
Description: Percentage of participants with throat pain. Throat pain severity will be assessed using a standard 0-10 scale, with higher scores indicating greater pain.
Time Frame: Up to 1 year
Population: Treated patients experiencing throat pain.
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 96 [87.9 to 98.6]

16. Secondary Outcome: Narcotic Analgesia Use
Description: Percentage of patients using narcotic analgesia during treatment.
Time Frame: Up to 2 years
Population: Treated patients that used a narcotic analgesic.
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 47
percentage of participants | 55 [41 to 69]

17. Secondary Outcome: Breaks in Chemoradiotherapy
Description: Mean number of breaks in chemoradiotherapy with LLLT use.
Time Frame: Up to 2 years
Population: Treated patients that experienced breaks in chemoradiotherapy.
Measure: Mean (Standard Deviation); unit: events
Arm/Group | Low Level Laser Therapy
Number analyzed (Participants) | 38
events | 47.7368 (5.19191)

ADVERSE EVENTS:
Time Frame: Adverse Events monitored up to 24 months, All-Cause Mortality monitored up to 36 months
Description: Adverse Events: Grade 1 and Grade 2 events per CTCAE v4.0 Serious Adverse Events: Grade 3 and Grade 4 events per CTCAE v4.0
Arm/Group | Low Level Laser Therapy
All-Cause Mortality (participants affected / at risk) | 7/47
Serious Adverse Events (participants affected / at risk) | 18/47
Other Adverse Events (participants affected / at risk) | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Level Laser Therapy (N=47)
Oral Mucositis (Gastrointestinal disorders) | 11
dysphagia (Gastrointestinal disorders) | 18
dry mouth (Gastrointestinal disorders) | 1
dermatitis (Injury, poisoning and procedural complications) | 2
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Low Level Laser Therapy (N=47)
Oral Mucositis (Gastrointestinal disorders) | 34
dysphagia (Gastrointestinal disorders) | 29
dry mouth (Gastrointestinal disorders) | 46
dysgeusia (Nervous system disorders) | 47
dermatitis (Injury, poisoning and procedural complications) | 45
oral pain (Gastrointestinal disorders) | 44
sore throat (Respiratory, thoracic and mediastinal disorders) | 45

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-12-03): https://cdn.clinicaltrials.gov/large-docs/92/NCT02682992/Prot_SAP_000.pdf